CLINICAL TRIAL: NCT06422949
Title: A Study on the Efficacy and Safety of HILOTERM® Device for the Prevention of Chemotherapy-induced Peripheral Neuropathy in Early Breast Cancer Patients
Brief Title: Efficacy and Safety of HILOTERM® Device for the Prevention of Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IEO 1974
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer; Neuropathy;Peripheral
Keywords: Early stage breast cancer; Paclitaxel; Chemotherapy-induced peripheral neuropathy
MeSH Terms: conditions — Breast Neoplasms; Neuritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hilotherm® Cooling treatment (Experimental): Cooling treatment with Hilotherm® at hands and feet level
  Interventions: Device: Hilotherm® Cooling treatment

INTERVENTIONS:
Device: Hilotherm® Cooling treatment — Patient will receive cooling treatment with Hilotherm® at hands and feet level from half an hour before taxol treatment start until half an hour after treatment end

SUMMARY:
Taxol is a very effective drug in breast cancer, but it can cause peripheral neuropathy (PN). This toxicity is often dose-limiting. Symptoms of PN usually improve after taxol discontinuation, but >80% of affected women experience symptoms 1-3 years after treatment stop. The intensity, the duration and the type of symptoms related to PN are very different and they can strongly interfere with patients' quality of life.

The application of cold to the hands and feet seems to be able to reduce the incidence of PN. Hilotherm® is a machine that allows to cool hands and feet. The aim of this study is to verify whether the use of Hilotherm® is able to reduce the incidence of moderate and severe PN and to evaluate the tolerability of Hilotherm® and its impact on quality of life.

DETAILED DESCRIPTION:
Taxol is a very effective drug in breast cancer, but it can cause peripheral neuropathy (PN), that is damage to the nerves of the hands and feet. This toxicity can begin a few days to months after starting taxol treatment and is often dose-limiting.

Symptoms of chemotherapy-induced peripheral neuropathy (CIPN) usually improve after taxol discontinuation, but >80% of affected women experience symptoms 1-3 years after treatment stop. The intensity, the duration and the type of symptoms related to PN are very different and they range from mild and transient symptoms to more severe and persistent symptoms. These symptoms can strongly interfere with patients' quality of life and can create difficulties in carrying out activities of daily living.

Despite numerous pharmacological approaches, no substance has proven capable of counteracting the onset of PN in patients eligible to receive chemotherapy with taxol. Some clinical studies have shown that the application of cold to the hands and feet is able to reduce the incidence of PN because the cold-induced constriction of the vessels leads to a reduction of blood flow and consequently to a reduced inflow of drug at the level of the hands and feet.

Hilotherm® is a machine that allows to keep hands and feet at a constant temperature of 10°C. The aim of this study is to verify whether the use of Hilotherm® is able to reduce the incidence of moderate and severe PN and to evaluate the tolerability of Hilotherm® and its impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women > 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Radically operated infiltrating breast cancer, pT1-T3, pN0-2, M0
* Candidate to adjuvant chemotherapy that includes weekly paclitaxel 80 mg/m2 intravenous for 12 weeks [either following anthracyclines and/or in association with trastuzumab]
* Negative pregnancy test at baseline (in fertile women)
* Willing and able to sign informed consent for protocol treatment

Exclusion Criteria:

* Evidence of metastatic disease (M1)
* pT4 and/or pN3
* Previous or concomitant malignancy of any other type
* Previous treatment with chemotherapy, hormonal therapy or an investigational drug for any type of malignancy
* Plans to use a chemotherapy regimen other than those specified in the inclusion criteria
* Any serious concurrent infection or any clinically significant medical illness (in particular clinically significant liver disease, clinically significant renal dysfunction, clinically significant cardiovascular disease, uncontrolled infections) which would jeopardize the ability of the patient to complete the planned therapy and follow-up
* Pre-existing motor or sensory neuropathy of any grade, for any reason
* Participation in any other clinical investigation or exposure to other investigational agents, drugs, device or procedure that may cause PN
* History of Raynaud phenomenon, either primary or secondary to autoimmune or connective tissue diseases such as systemic lupus erythematous, scleroderma, Buerger disease, Sjögren syndrome, rheumatoid arthritis, occlusive vascular disease, such as atherosclerosis, polymyositis, cold agglutinin disease or cryoglobulinemia, thyroid disorders, pulmonary hypertension
* Cold urticaria / cold contact urticaria
* Severe arterial disease
* Trophic tissue lesions
* Diabetes mellitus
* Alcohol abuse
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to the components of Hilotherm Chemo care device
* Simultaneous use of Dignicap system to prevent hair loss from chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Overall incidence of grade 2 or 3 CIPN | 12 months
  Severity of PN evaluated using the CTCAE scale, version 5

SECONDARY OUTCOMES:
Incidence of withdrawal from Hilotherapy | 12 weeks
  Number of patients withdrawing Hilotherapy due to cold intolerance
Patients' physical, psychological and social functions evaluation | 12 months
  Collection of EORTC QLQ-C30 [European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire] (minimum value: 1, maximum value: 4 - higher scores mean a worse outcome)
Side effects impact evaluation | 12 months
  Collection of EORTC-BR23 [European Organization for Research and Treatment of Cancer - Breast Cancer specific Module] (minimum value: 1, maximum value: 4 - higher scores mean a worse outcome)
Pain assessment | 12 months
  Collection of Brief Pain Inventory (BPI) questionnaire (minimum value: 0, maximum value: 10 - higher scores mean a worse outcome)
Technology acceptance and perception evaluation | 12 months
  Collection of Technology Acceptance Model Questionnaire (minimum value: 1, maximum value: 7 - higher scores mean a lower agreement with the statement)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Dellapasqua, MD, Principal Investigator — European Istitute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy